CLINICAL TRIAL: NCT04670341
Title: Quality Improvement of Saliva by Chewing Tapioca Pearls in Bubble Tea Drinks
Brief Title: The Effect of Chewing the Tapioca Pearls in Bubble Tea Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Juni Handajani, Quality improvement of saliva by chewing tapioca pearls in bubble tea drinks, Gadjah Mada University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FKGUGM1
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Saliva
Keywords: bubble tea; salivary C-reactive protein; salivary calcium

STUDY DESIGN:
Intervention Model Description: In the first week of the experiment, subject chewing tapioca pearl inthe bubble tea. In the second week, the same subjects drink tea without chewing tapioca pearl
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- chewing tapioca pearls in the bubble tea drinks (Experimental): In the first week, the subjects drink as much as 100 ml of bubble tea over a span of 5 minutes once a day for 3 days
  Interventions: Other: chewing tapioca pearls in bubble tea drinks
- drink tea without chewing tapioca pearls (Placebo Comparator): In the second week, the subjects drink tea without tapioca pearls as much as 100 ml for 5 minutes per day for 3 days.
  Interventions: Other: drink tea without chewing tapioca pearls

INTERVENTIONS:
Other: chewing tapioca pearls in bubble tea drinks — Saliva was collected on the first day before bubble tea consumption (pretest) and on the third day after bubble tea consumption (posttest); collection was conducted in the morning (09:00 a.m.-12.00 p.m.).
  Arms: chewing tapioca pearls in the bubble tea drinks
Other: drink tea without chewing tapioca pearls — Saliva was collected on the first day before drink tea without tapioca pearl (pretest) and on the third day after tea consumption (posttest); collection was conducted in the morning (09:00 a.m.-12.00 p.m.).
  Arms: drink tea without chewing tapioca pearls

SUMMARY:
Bubble tea drinks contain tea and tapioca pearls. Chewing tapioca pearls in bubble tea drinks may increase salivary components. Because of its proteins, inorganic components, and enzymes, saliva plays an important role in the body's defense against bacteria and viruses. This study aims to analyze the effect of chewing the tapioca pearls in bubble tea drinks on salivary C-reactive protein (CRP) and calcium (Ca) levels.

DETAILED DESCRIPTION:
Sixty saliva samples were collected from 15 subjects. The inclusion criterion was 18-25 years of age. The exclusion criteria were receiving medication, using dentures, a history of dry mouth, smoking and systemic disease. In the first week of the experiment, subjects drank bubble tea as the intervention group. In the second week, the same subjects drank tea without pearls as the control group. Each subject drank the bubble tea for 5 minutes per day over 3 days. Saliva samples were collected on the first day before bubble tea consumption (pretest) and on the third day after tea consumption (posttest). Saliva collection was performed in the morning (09:00 a.m.-12:00 p.m.) for 1 minute. Salivary CRP levels were measured using an ELISA kit, and Ca levels were determined using a test kit.

ELIGIBILITY:
Inclusion Criteria:

* good Oral Hygiene Index-Simplified (OHI-S) score

Exclusion Criteria:

* taking medication
* a history of dry mouth
* smoking
* systemic disease

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Salivary C-reactive protein (CRP) level | 3 days
  Salivary CRP level was measured on the first day before chewing tapioca peals in the bubble tea drinks and drink tea. Salivary CRP level was measured on the third day after drink bubble tea and tea without tapioca pearls

SECONDARY OUTCOMES:
Calcium (Ca) level | 3 days
  Ca level was measured on the first day before chewing tapioca peals in the bubble tea drinks and drink tea. Ca level was measured on the third day after drink bubble tea and tea without tapioca pearls

CONTACTS AND LOCATIONS:
Overall Officials: Juni Handajani, PhD, Principal Investigator — Faculty of Dentistry, Universitas Gadjah Mada
Locations (1):
- Faculty of Dentistry, Universitas Gadjah Mada, Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handajani J, Kusumajati D, Fathiyah H, Susilowati H, Tandelilin RTC. Quality improvement of saliva by chewing tapioca pearls in bubble tea drinks: a randomized experimental trial: (Study on salivary C-reactive protein (CRP) and calcium (Ca) levels). F1000Res. 2021 Feb 1;10:56. doi: 10.12688/f1000research.28028.2. eCollection 2021. PMID 35387272
- See also: Elevated salivary C-reactive protein levels are associated with active and passive smoking in healthy youth: A pilot study — https://doi.org/10.1186/1476-9255-8-37